CLINICAL TRIAL: NCT03395977
Title: Differential Effects of Uric Acid and Xanthine Oxidoreductase on Endothelial Function and Oxydative Stress
Brief Title: Uric Acid Effects on Endothelium and Oxydative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Fonds Erasme (Unknown); Fonds National de la Recherche Scientifique (Other)
Responsible Party: Principal Investigator, Benjamin De Becker, Investigator, Clinical Research, Erasme University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 30309647
Record Dates: First submitted 2017-12-29; First posted 2018-01-10 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Oxidative Stress; Endothelial Function; Cardiovascular System; Hypertension
Keywords: uric acid; xanthin oxydoreductase; febuxostat; uricase
MeSH Terms: conditions — Hypertension | interventions — Febuxostat; rasburicase

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, placebo-controlled, double-blinded and 3 ways cross-over study.
  Three populations : healthy male subjects under 40 y [1] ; healthy male and female participants between 40 and 65 years [2] and subjects with hypertension [3]. Minimum 15 participants in each group are needed.
  The populations 2 and 3 will be studied together with subgroups analyses of the results for the status of hypertension, of treatment, age and gender.
  For 5 subjects in each group, we will perform a fourth session with Placebo PO and Rasburicase IV. That session will be non-randomized and blinded only for the subject.
Who Masked: Participant, Investigator
Masking Description: Febuxostat and Rasburicase will be prepared by an independant pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebos PO and IV (Placebo Comparator): PO : per os IV : intraveinously
  Interventions: Drug: Placebos
- Febuxostat PO and Placebo IV (Experimental): 240 mg a day for 3 days
  Interventions: Drug: Placebos; Drug: Febuxostat
- Febuxostat PO And Rasburicase IV (Experimental): Febuxostat : 240 mg a day for 3 days. Uricase : 3 mg once.
  Interventions: Drug: Febuxostat; Drug: Rasburicase
- Placebo PO And Rasburicase IV (Experimental): Placebo : for 3 days. Uricase : 3 mg once.
  Interventions: Drug: Placebos; Drug: Rasburicase

INTERVENTIONS:
Drug: Placebos — Lactose placebo for pills and saline for perfusion.
  Other Names: Placebo
  Arms: Febuxostat PO and Placebo IV; Placebo PO And Rasburicase IV; Placebos PO and IV
Drug: Febuxostat — Febuxostat tablet.
  Other Names: Adenuric
  Arms: Febuxostat PO And Rasburicase IV; Febuxostat PO and Placebo IV
Drug: Rasburicase — Rasburicase injectable solution.
  Other Names: Fasturtec
  Arms: Febuxostat PO And Rasburicase IV; Placebo PO And Rasburicase IV

SUMMARY:
Cardiovascular disease is the leading cause of mortality worldwide. Endothelial dysfunction (ED) is the main mechanism which leads to atherosclerosis, where the balance between pro and antioxidant factors results in a decreased nitric oxide (NO) bioavailability. Xanthine OxidoReductase (XOR) is one of the main generators of reactive oxygen species (ROS). Uric acid (UA), a major antioxidant in human plasma and end product of purine metabolism, is associated with cardiovascular diseases since many years; however the precise mechanisms which relate UA to ED are still not well understood.

The purpose of this study is to unravel the XOR and UA pathways involved in ED. Three groups of participants (young (< 40 y) male healthy participants [1] ; male and female helthy participants (40 to 65 y) [2] and patients with primary hypertension [3]) will be exposed to febuxostat (a strong and selective XOR inhibitor), or recombinant uricase (which oxidizes UA into allantoin) to vary UA levels and concomitantly control for confounding changes in XOR activity. Oxidative stress will be estimated by several markers. Endothelial function will be assessed by a laser Doppler imager in the presence of hyperthermia and endothelium stimulators. This study is specifically designed to untie the respective effects of UA and XOR pathways on oxidative stress and endothelial function in humans.

The investigators will test the following hypothesis:

1. An extremely low level of uric acid after uricase administration induces endothelial dysfunction and oxydative stress,
2. A specific XO inhibitor limits unfavourable effects of the serum UA reduction elicited by uricase administration,
3. Endothelial function and oxydative stress are further improved with febuxostat as compared to placebo,
4. All these observations are more marked in hypertensives then in older participants than in young healthy subjects.

DETAILED DESCRIPTION:
The goals of the research protocol are to clearly untie the respective roles of uric acid (UA) and xanthine oxidoreductase (XOR) pathways on endothelial function and oxidative stress in humans.

UA represents the end-product of purine metabolism due to the loss of uricase 15 million years ago in humans. The selective advantage of this mutation could be the strong antioxidant effect of UA (which represents more than 60% of the antioxidant plasmatic capacity). Many recent epidemiological studies have showed a J-shape association between UA levels and cardiovascular risk. An UA level lower than 3 mg/dl could be damageable due to the loss of the antioxidant properties of UA. In contrast, hyperuricemia is associated with an increased inflammation, insulin resistance, ED, platelet aggregation, left ventricle hypertrophy, arterial vasodilatation impairment, aortic stiffness and intima-media thickness. However, the association between UA and cardiovascular disease remains controversial because whether UA is an independent risk factor for these illnesses is unclear.

Interventional studies:

Because the above-mentioned associations do not prove causation, several authors designed interventional studies with the purpose to modify UA levels and determine if this affected endothelial function and oxidative stress. The main limitation of these studies is that they were unable to untie the effects of the synthesis of UA, of UA itself and of the activity of XOR, on ROS production and endothelial function in humans.

This is because:

1. serum UA is a powerful plasmatic antioxidant,
2. but transformation of hypoxanthine to xanthine and xanthine to UA by XO generates intracellular ROS,
3. moreover, in endothelial cells, UA reduces NO bioavailability by many ways (L-arginine blockade and degradation, increased superoxide anion production, NOS inhibition, reduced NOS genes expression and direct NO scavenging),
4. in addition, UA forms crystals in the endothelium wall which create a pro-inflammatory and thrombotic state, increases smooth muscle cells proliferation and also insulin resistance and inflammation in adipocytes,
5. finally, and most importantly, XO is inhibited by physiologic levels of UA (which acts as an uncompetitive XO inhibitor).

In summary, the present protocol aims at testing the following hypothesis:

1. Experimental serum UA variations are correlated with endothelial function and oxydative stress markers : an extremely low level after uricase administration induces ED and oxydative stress,
2. A specific XO inhibitor (FX) limits unfavourable effects of the serum UA reduction elicited by uricase administration, since this will hamper the feedback activation of XO by a low UA level,
3. Endothelial function and oxydative stress are further improved with FX as compared to placebo, because the first experimental condition results in a XO blockade,
4. All these observations are more marked in hypertensive patients then in older participants than in young healthy subjects.

Data collection

Data collection from the participants will be collected informatically through a case report form. The names and personnal data from the patients will be kept in a secret place or in a password-protected file. All the data will be destroyed at the end of the study (including blood and urine samples).

Statistical analysis

Statistical analysis will be performed using SPSS. Baseline characteristics will be compared using a Student t test. Two-way repeated-measures ANOVAs will be used to detect significant changes between sessions and groups. Statistical significance is assumed when p is <0.05. Sample size is not possible due to the lack of data of the effect of acute hypouricemia. We estimate a minimum of 15 participants in each group.

Specific test will be used for non gaussian variables. Correlation test will be used if necessary according the results of the first test.

Placebo-corrected values and comparisons of the delta will be used too.

Subgroups analyses will be performed for the study of population 2 and 3 (enrolled together).

ELIGIBILITY:
Phase 1 :

Inclusion Criteria:

* Age between 18 and 40 years
* Male
* Healthy volunteers
* Non smoker for at least 6 months
* Uric acid level in normal range (normouricemic group)

Exclusion Criteria:

* Any diseases of one of the following systems: cardiovascular, digestive, hormonal, urinary, pulmonary, rheumatic or immune.
* Smoker, alcoholic
* Participants should not take any chronic medicine nor vitamins or other antioxidants.
* A G6PD deficit will be excluded as this is a contraindication to uricase administration (hemolytic anemia).

Phase 2 :

Inclusion Criteria:

* Age between 40 and 65 years
* Male or female (menopaused)
* Healthy volunteers
* Non smoker for at least 6 months
* Uric acid level in normal range (normouricemic group)

Exclusion Criteria:

* Any diseases of one of the following systems: cardiovascular, digestive, hormonal, urinary, pulmonary, rheumatic or immune.
* Smoker, alcoholic
* Participants should not take any chronic medicine nor vitamins or other antioxidants.
* A G6PD deficit will be excluded as this is a contraindication to uricase administration (hemolytic anemia).

Phase 3 :

Inclusion Criteria:

* Age between 40 and 65 years
* History of hypertension for more than 6 months
* Non smoker or smoke stopped for at least for 6 months

Exclusion Criteria:

* Acute coronary syndrome
* Heart failure (LVEJ < 40%)
* Diabetes
* Active smoking
* Gout
* Chronic kidney disease stage superior to 3a
* History of cerebrovascular thrombosis
* Cirrhosis
* Alcohol consumption more than 3 units/day
* Participants should not take any chronic medicine nor vitamins or other antioxidants.
* A G6PD deficit will be excluded as this is a contraindication to uricase administration (hemolytic anemia).

The populations of phases 2 and 3 will be enrolled and studied together with subgroups analyses of the results for the status of hypertension, of treatment, age and gender.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female for phases 2 and 3
Enrollment: 53 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Cutaneous perfusion by Laser Doppler (perfusion unit) | 24 hours after infusion of Uricase or Placebo
  Perfusion unit (Laser Doppler Imager + iontophoresis of (ACh and SNP and hyperemia with ou without L-NAME). Assessment of endothelial function.

SECONDARY OUTCOMES:
Change in Oxydative stress biomarkers from baseline to 30 min or 24 hours after infusion of Uricase or Placebo | Baseline, 30 minutes and 24 hours after infusion of Uricase or Placebo
Arterial stiffness | 24 hours after infusion of Uricase or Placebo
  Carotido-femoral and carotido-radial pulse wave velocity and pulse wave analysis
Blood pressure (mmHg) | 24 hours after infusion of Uricase or Placebo
  Beat-to-beat measurements with Finapres and manually
Cardiac output (l-min) | 24 hours after infusion of Uricase or Placebo
  Beat-to-beat measurements with Finapres
Change in enzymes activity | 30 min and 24 hours after infusion of Uricase or Placebo
  Xanthin oxydase activity
Change in enzymes expression | 30 min and 24 hours after infusion of Uricase or Placebo
  eNOS, NOX, XO we will incubate endothelial cells with plasma or serum from subjects. Then we will measure the sus-mentionned enzymes' expression.
Change in proteomic or metabolomic analysis | 30 min and 24 hours after infusion of Uricase or Placebo
  We will perform proteomics or metabolomics analysis directly on serum from participants and also on lysate of endothelial cells pre-incubated with plasma or serum from participants.
Change in renin-angiotensin activity | Baseline, 30 minutes and 24 hours after infusion of Uricase or Placebo
Change in urinary excretion of sodium | Baseline, 30 minutes and 24 hours after infusion of Uricase or Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Philippe van de Borne, Study Director — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgique, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Becker B, Hupkens E, Dewachter L, Coremans C, Delporte C, van Antwerpen P, Franck T, Zouaoui Boudjeltia K, Cullus P, van de Borne P. Acute effects of hypouricemia on endothelium, oxidative stress, and arterial stiffness: A randomized, double-blind, crossover study. Physiol Rep. 2021 Sep;9(17):e15018. doi: 10.14814/phy2.15018. PMID 34435469
- [Derived] De Becker B, Coremans C, Chaumont M, Delporte C, Van Antwerpen P, Franck T, Rousseau A, Zouaoui Boudjeltia K, Cullus P, van de Borne P. Severe Hypouricemia Impairs Endothelium-Dependent Vasodilatation and Reduces Blood Pressure in Healthy Young Men: A Randomized, Placebo-Controlled, and Crossover Study. J Am Heart Assoc. 2019 Dec 3;8(23):e013130. doi: 10.1161/JAHA.119.013130. Epub 2019 Nov 22. PMID 31752638